CLINICAL TRIAL: NCT02771704
Title: In Vivo Evaluation of the Antimicrobial Activity of Diamine Silver Fluoride and Potassium Iodide on Dentin Carious Lesions in Kuwaiti Subjects.
Brief Title: Diamine Silver Fluoride and Potassium Iodide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Maribasappa Karched, Assistant Professor, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KuwaitU
Record Dates: First submitted 2016-05-01; First posted 2016-05-13 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Dentine Caries
MeSH Terms: interventions — silver diamine fluoride; Potassium Iodide; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Silver diamine fluoride (Experimental): Intervention: Silver diamine fluoride will be applied in vivo on carious dentine lesions
  Interventions: Other: Silver Diamine fluoride
- Potassium iodide (Experimental): Potassium iodide will be applied in vivo on carious dentine lesions.
  Interventions: Other: Potassium iodide
- Chlorhexidine (Experimental): Chlorhexidine will be applied in vivo on carious dentine lesions
  Interventions: Other: Chlorhexidine
- Silver diamine fluoride+Potassium iodide (Experimental): Silver diamine fluoride and potassium iodide mixture will be applied in vivo on carious dentine lesions
  Interventions: Other: Silver diamine fluoride and potassium iodide
- Saline (Experimental): Sterile physiological saline will be applied in vivo on carious dentine lesions
  Interventions: Other: Physiological saline

INTERVENTIONS:
Other: Silver Diamine fluoride
  Arms: Silver diamine fluoride
Other: Potassium iodide
  Arms: Potassium iodide
Other: Chlorhexidine
  Arms: Chlorhexidine
Other: Silver diamine fluoride and potassium iodide
  Arms: Silver diamine fluoride+Potassium iodide
Other: Physiological saline
  Arms: Saline

SUMMARY:
Dental caries is an infectious disease mediated by a consortium of microbes in the oral cavity. The disease is characterized by demineralization of the tooth, if untreated, it leads to cavitation, discomfort, pain and eventual tooth loss. Frequently, complete caries removal of dentine carious lesions leads to exposure of the pulp affecting its vitality. Therefore, it is crucial that vitality of the teeth is preserved causing little damage to the pulp. Different approaches have been used to reduce or eliminate microorganisms underneath the restorations. Chlorhexidine has a strong antibacterial effect, particularly on planktonic bacteria. Its effect on bacterial biofilms is compromised, however The objective of this study is to examine the in vivo effect of diamine silver fluoride, potassium iodide and their mixture on bacteria present in deep carious lesions. Dentine samples from 5 carious lesions from each of 5 patients before and after treatment with test agents will be collected in pre-reduced sterile Ringer's solution and processed for microbiological evaluation. The samples after serial dilution and plating will be incubated in aerobic, anaerobic and CO2 atmosphere for 2-5 days. Colony forming units will be enumerated and the effect of antibacterial agents in question on the bacterial viability in carious lesions will be assessed.

DETAILED DESCRIPTION:
Study subjects:

Study subjects (n=5) will be recruited from the pool of patients attending Kuwait University Dental Clinic. Informed written consent will be obtained from all subjects. An approval for using human subjects in the study will be obtained from the Ethics Committee of HSC, Kuwait University.

Inclusion criteria:

* Patient is able to give informed consent
* Tooth with moderate size caries lesions, penetrate through ½ of dentine thickness
* Suitable for the placement of a Vitrabond lining
* Restoration is part of a current and approved treatment plan

Exclusion criteria:

* Patient is unable to give informed consent
* Teeth had received temporary restoration
* Isolation with rubber dam is not possible
* Cavity preparation was contaminated due to gingival bleeding

Clinical protocol The cavity will be restored using materials and methods which has been approved by KUDC, the use of Vitrabond liner is essential as part of this study.

Sample collection: Decayed dentine will be removed by using a sterile dental excavator and collected into a sterile microfuge tubes for microbiological analyses before treatment. Using a dental three-in-one air syringe, the tooth surface will then be cleaned using sterile distilled water and dried for 4 sec. The lesions will be treated with Silver diamine fluoride, potassium iodide or their mixture (SDI Ltd., Melbourne, Australia), a product made of silver diamine fluoride (38% w/v) and a saturated solution of potassium iodide and an oxalic acid based product which contains oxalic acid, potassium salt and water. In parallel, Chlorhexidine and sterile saline will be used as control treatment agents. After treatment, dentin samples will be collected using a sterile dental excavator. Followed by excavation, all three treatment agents will be applied for 30 sec and samples will be collected once again after the treatment.

Microbiological analysis: The samples after collection will be immediately placed on ice and brought within 30 min to the Oral Microbiology lab at the Faculty of Dentistry. Standard protocols will be followed for microbiological culture. Samples collected in pre-weighed sterile microfuge tubes will be weighed again to determine weight of the dentine material. Dentin samples will then be suspended in sterile pre-reduced Ringer's solution.. After vigorously vortexing for 1 min at maximal setting, samples will be 10-fold serially diluted up to 10-6 in Ringer's solution. Initially in pilot experiments, samples will be cultured on different media in CO2, aerobic and anaerobic conditions. One hundred microliter from each dilution will be spread in two sets in duplicate on the following media and incubated:

1. Brucella agar plates supplemented with 5% sheep blood for total viable bacterial count. Plates will then be incubated in 5% CO2 and anaerobic atmosphere (85% Nitrogen, 10% Hydrogen and 5% CO2) at 37 C for 2 days. Anaerobic condition in the jars will be monitored using RT Anaero-Indicator (Mitsubishi Gas Chemical Company Inc., Japan).
2. Mitis salivarius agar (Difco) for Streptococcus spp. count; incubation in 5% CO2 in air at 37 C for 2 days.
3. Mitis salivarius agar supplemented with 20% sucrose, bacitracin (0.2 units/ml) and 1% potassium tellurite for Streptococcus mutans count; incubation at 37 C in 5% CO2 in air for 2 days.

After incubation plates will be removed from the jars and colony forming units (CFU) will be enumerated from appropriate dilutions. CFUs will be calculated per milligram of the sample taken . All experiments will be performed in triplicate.

Statistical analysis:

At least three independent experiments, each sample run in duplicates, will be performed. ANOVA will be used for comparing bacterial counts before and after the application of the treatment agent. testing the effect of the treatment agent. Mann-Whitney U test will be used to compare CFU counts between test and control groups. A p value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be able to give informed consent.
* had at least 5 teeth with moderate size caries lesions (for 5 treatments), to be exact with the lesion size.
* the carious lesion should at least penetrate to the inner ½ of dentine thickness.
* the lesion should be suitable for the placement of a Vitrabond lining of 0.5-1.0 mm
* permanent restoration should be a part of a current and approved treatment plan

Exclusion Criteria:

* Inability of the patient to give informed consent.
* teeth had received temporary restoration
* isolation with rubber dam is not possible.
* if cavity preparation was contaminated due to gingival bleeding

All patients were placed under a follow up system for the purpose of addressing any complaints that might result from the sampling procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
antibacterial activity measured by total viable counts after treatment | Through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maribasappa Karched, PhD, Principal Investigator — Kuwait University

REFERENCES:
- [Background] Jouseimies-Somer H, Summanen P, Citron DM, Baron EJ, Wexler HM, Finegold S, (2002) Anaerobic Bacteriology Manual, Wadsworth-KTL.
- [Background] Emilson CG, Bratthall D. Growth of Streptococcus mutans on various selective media. J Clin Microbiol. 1976 Jul;4(1):95-8. doi: 10.1128/jcm.4.1.95-98.1976. PMID 956364